CLINICAL TRIAL: NCT01461642
Title: E-support for Healthcare Processes - ASTHMA
Acronym: E-ASTHMA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Collaborators: University of Primorska (Other)
Responsible Party: Principal Investigator, Mateja Marc Malovrh, MD, PhD, The University Clinic of Pulmonary and Allergic Diseases Golnik
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: L7 - 3653 - ASTHMA
Record Dates: First submitted 2011-10-26; First posted 2011-10-28 (Estimated); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Asthma
Keywords: Asthma; ICT Support; ACT; PEF
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Asthma - ICT support. (Experimental)
  Interventions: Other: Self management asthma plan indorsment.
- Asthma, comparator - no ICT support (No Intervention)

INTERVENTIONS:
Other: Self management asthma plan indorsment. — Subjects adherence to asthma self management plan will be monitored through web-based support.
  Arms: Asthma - ICT support.

SUMMARY:
The purpose of the study is to establish and clinically evaluate a new approach to treating asthma by using information and communication technologies (ICT). A mobile environment, and organizational interventions to improve the process of an integrated treatment of people with asthma will be identified, developed, introduced and clinically evaluated.

DETAILED DESCRIPTION:
A mobile environment to improve the process of an integrated treatment of people with asthma will be identified, developed, introduced and clinically evaluated. The study will include 120 patients diagnosed with asthma that is poorly managed. The study will use the ACT (Asthma Control Test) questionnaire and an evaluation questionnaire that will cover issues regarding the satisfaction of subjects with asthma care offered. Subjects with a PEF meter, will be able to enter the value of PEF (Peak Expiratory Flow).

In addition to this, users can enter values (1) physical activity (type, duration, intensity), and (2) food (type, quantity).

ELIGIBILITY:
Inclusion Criteria:

* ACT points <19
* Daily symptoms> = 2 days/week
* Night symptoms> = 1 night/week
* Rescue medication > 2days/week
* At least one asthma exacerbation in the past year, but not in the last month, which was treated with oral glucocorticoid

Exclusion Criteria:

* Worsening of asthma in the last 4 weeks (treated with oral corticosteroids)
* Age >70 or <18 years
* Significant co-morbidity
* Does not own or know how to handle a mobile phone
* No internet access
* Not able to perform a PEF measurment
* Not able to use inhalor

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10; Primary Completion 2016-11-14 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Number of exacerbations. | 1 year
  Number of exacerbations per year.

CONTACTS AND LOCATIONS:
Locations (1):
- University Clinic of Pulmonary and Allergic Disease, Golnik, Slovenia